CLINICAL TRIAL: NCT03211338
Title: Inflammation and Cell Maturation in Preterm Delivery Placentas - in Vitro and in Vivo Effect of Progesterone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HYMC-0061-17
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Obstetric Labor, Premature
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Culture Techniques; Progesterone; Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Preterm labor placentas and progesterone (Active Comparator): IMC cells taken from preterm labor placentas after delivery will be cultured with progesterone and will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture with progesterone
- Term labor placentas and progesterone (Active Comparator): IMC cells taken from term labor placentas after delivery will be cultured with progesterone and will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture with progesterone
- Preterm labor placentas without progesterone (Active Comparator): IMC cells taken from preterm labor placentas after delivery will be cultured without progesterone and will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture without progesterone
- Term labor placentas without progesterone (Active Comparator): IMC cells taken from term labor placentas after delivery will be cultured without progesterone and will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture without progesterone
- Term placentas from progesterone treated pregnancies (Active Comparator): IMC cells taken from term labor placentas from women that were treated with progesterone during pregnancy will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture with growth factors
- Preterm placentas from progesterone treated pregnancies (Active Comparator): IMC cells taken from preterm labor placentas from women that were treated with progesterone during pregnancy will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture with growth factors
- Term placentas not treated with progesterone in pregnancy (Active Comparator): IMC cells taken from term placentas from women who were not treated with progesterone during pregnancy will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture with growth factors
- Preterm placentas not treated with progesterone in pregnancy (Active Comparator): IMC cells taken from preterm placentas from women who were not treated with progesterone during pregnancy will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture with growth factors
- Term postpartum blood samples with progesterone (Active Comparator): CD-14+ monocyte cells taken from women delivering at term will be cultured with progesterone and will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture with progesterone
- Preterm postpartum blood samples with progesterone (Active Comparator): CD-14+ monocyte cells taken from women delivering preterm will be cultured with progesterone and will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture with progesterone
- Term postpartum blood samples without progesterone (Active Comparator): CD-14+ monocyte cells taken from women delivering at term will be cultured without progesterone and will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture without progesterone
- Preterm postpartum blood samples without progesterone (Active Comparator): CD-14+ monocyte cells taken from women delivering preterm will be cultured without progesterone and will be analyzed for inflammation characteristics and maturation into DC cells.
  Interventions: Biological: Culture without progesterone

INTERVENTIONS:
Biological: Culture with progesterone — Progesterone, a steroid hormone will be cultured with placental IMC cells or peripheral blood CD14+ monocyte cells
  Arms: Preterm labor placentas and progesterone; Preterm postpartum blood samples with progesterone; Term labor placentas and progesterone; Term postpartum blood samples with progesterone
Biological: Culture without progesterone — Culture of placental IMC cells or peripheral blood CD14+ monocyte cells without progesterone
  Arms: Preterm labor placentas without progesterone; Preterm postpartum blood samples without progesterone; Term labor placentas without progesterone; Term postpartum blood samples without progesterone
Biological: Culture with growth factors — Culture of placental IMC cells with growth hormones only and analysis
  Arms: Preterm placentas from progesterone treated pregnancies; Preterm placentas not treated with progesterone in pregnancy; Term placentas from progesterone treated pregnancies; Term placentas not treated with progesterone in pregnancy

SUMMARY:
The aim of this study is to investigate the In Vitro and In Vivo effect of progesterone on immature myeloid cells (IMC), inflammation characteristics and maturation into dendritic cells (DC).

ELIGIBILITY:
Inclusion Criteria:

* Placentas from term and preterm deliveries
* Singleton pregnancy
* Consent to participate

Exclusion Criteria:

* Pregnancies with obstetric complications
* Multiple gestation
* Maternal illness or fetal malformation known pre-delivery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Inflammation characteristic effects of progesterone on preterm and term placentas | One year
  Differences observed in cytokine profiles of IMC cells from term and preterm placentas cultured with and without progesterone
Maturation effects of progesterone on preterm and term placentas | One year
  Differences observed in maturation of IMC cells into DC cells in term and preterm placentas

CONTACTS AND LOCATIONS:
Overall Officials: Rinat Gabbay-Benziv, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No